CLINICAL TRIAL: NCT06855199
Title: INVESTIGATION OF THE CORRELATION OF BLOCK SUCCESS WITH GALVANIC SKIN RESPONSE IN PEDIATRIC SURGERY CASES PERFORMED UNDER CAUDAL EPIDURAL BLOCK ANESTHESIA
Brief Title: CAUDAL EPIDURAL BLOCK IN PEDIATRIC SURGERY CASES
Status: Recruiting | Type: Observational
Sponsor: Cigdem Demirci (Other)
Collaborators: sivas devlet hastanesi (Other); Adiyaman University Research Hospital (Other)
Responsible Party: Sponsor-Investigator, Cigdem Demirci, doctor, sivas devlet hastanesi
Organization: sivas devlet hastanesi (Other)
Other Study IDs: SDH-AR-CD-01
Record Dates: First submitted 2024-11-28; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Patient
Keywords: GALVANİC SKİN RESPONSE; PEDIATRIC PATIENT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Caudal epidural anesthesia was reported as the first epidural anesthesia technique in 1933, but its use began to become widespread after the 1960s (1). The procedure is reliable, easy to perform, the incidence of complications is low, and the total complication rate is 1.5/1000; Serious complications occur at a rate of 1/40000. There are many methods to demonstrate the success of caudal epidural block. Some of the common traditional methods are changes in mean arterial pressure and heart rate. These methods are sometimes not objective and take time. In this study, we will examine the block success in pediatric patients who underwent caudal epidural block, which is applied in our hospital, whether the Galvanic skin response measured with a finger probe, other than traditional methods, correlates with the block success, and whether it shows faster block success compared to other traditional methods.

DETAILED DESCRIPTION:
A successful caudal epidural block can provide safe, effective regional anesthesia. (4). The overall failure rate of caudal epidural block in pediatric patients is approximately 4%, depending on the anatomical and developmental abnormalities of the caudal canal (5,6). Therefore, reliable and rapid evaluation of a successful caudal epidural block is important to optimize anesthesia management in pediatric patients. Evaluating the success of caudal epidural block with traditional methods such as mean arterial pressure (MAP) and heart rate (HR) does not give completely objective results and takes time. Galvanic Skin Response (GSR) is a parameter that shows sweat gland function related to the autonomic nervous system. Physically, the galvanic skin response is the change in the electrical structure of the skin in response to various stimuli (7).Changes in tension measured from the skin surface are recorded. The relaxation and calming response accompanies an increase in skin resistance, while the fight response accompanies a decrease in skin resistance. In general, low conductivity is a sign of relaxation. High conductivity is a sign of emotional, mental or physical arousal (8). Galvanic Skin Response (GSR) evaluation is a non-invasive measurement that allows us to observe skin resistance changes with two probes attached to the fingertip. The aim of this study is to evaluate whether using Galvanic skin response (GSR) values measured with a finger probe will detect the success of caudal epidural block more quickly than other traditional methods in pediatric patients who underwent surgery with caudal epidural block.

ELIGIBILITY:
Inclusion Criteria:

* lower abdominal/urogenital/lower extremity surgery
* Patients with ASA1-2

Exclusion Criteria:

* Those with neuromuscular disease
* PATIENTS WITH ASA3-4
* patients with cerebral palsy
* patients in mental reter

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: PEDIATRIC GROUP BETWEEN 1-6 YEARS
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of block success in patients undergoing caudal epidural block | After the caudal block is performed, it will be monitored for 20 minutes.
  Evaluation of block success in patients undergoing caudal epidural block

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas State Hospital, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No